CLINICAL TRIAL: NCT04962867
Title: Multicenter Investigator-initiated Phase II Trial of E7090 in Patients With Advanced or Recurrent Solid Tumor With Fibroblast Growth Factor Receptor (FGFR) Gene Alteration (FORTUNE Trial)
Brief Title: NCCH2006/MK010 Trial (FORTUNE Trial)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Center, Japan (Other Government)
Collaborators: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCH2006/MK010
Record Dates: First submitted 2021-07-12; First posted 2021-07-15 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Advanced or Recurrent Solid Tumors; FGFR Gene Alterations
Keywords: E7090; Solid tumor; Fibroblast Growth Factor Receptor (FGFR); FGFR inhibitor
MeSH Terms: conditions — Acrocephalosyndactylia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: E7090 — 140 mg of E7090 is orally administered once daily.

SUMMARY:
This is a single-arm, open-label, multicenter, investigator-initiated Phase 2 trial to evaluate the efficacy and safety of E7090 in patients with advanced or recurrent solid tumors harboring FGFR genetic alterations (including fusion, mutation, amplification).

ELIGIBILITY:
Inclusion Criteria:

1. Participants with histologically or cytologically confirmed metastatic, unresectable, or recurrent solid tumor who agree to provide an archival tumor sample, a residual biopsy sample, or a fresh tumor biopsy sample
2. Ineffective to or intolerant to initial treatment, or for which standard treatment is no longer available
3. Participants with an FGFR gene alteration detected by NGS panel, who fall under one of the categories of groups A to C and E defined as below

   Group A: FGFR1-3 fusion

   Group B and E: FGFR1-3 specific activating mutations as below;

   FGFR1: P150S, T340M, R445W, N546K, K656E

   FGFR2: C62Y, A67V, N82K, D101Y, E160K, E163K, M186T, R203H, R210Q, Q212K, R251Q, S252W, P253R, P253L, A264T, W290C, K310R, Y328N, G364E, Y375C, C382R, A389T, V392A, R399Q, H416R, I422V, H544Q, N549H, N549K, N549D, N549S, L560F, K659E, K659N, R664W, E718K, S791T

   FGFR3: G380E, G380R, A391E, K650T, K650E, K650Q, K650N

   Group C: FGFR1-3 activating mutation not applicable to group B, or FGFR1, 2 gene amplification
4. For Group D, participants with cholangiocarcinoma who have previously received a selective FGFR inhibitor other than E7090 and have demonstrated progressive disease or resistance
5. Karnofsky Performance Status (KPS) >= 70 for patients with primary CNS tumors. Performance Status (ECOG) 0-1 for patients with non-primary CNS tumors
6. For patients with non-primary CNS tumors, they have at least 1 lesion of >= 10 millimeter (mm) in the longest diameter for a non-lymph node or >= 15 mm in the short-axis diameter for a lymph node that is considered as serially measurable according to RECIST v1.1 using computerized tomography or magnetic resonance imaging (CT or MRI) within 28 days of enrollment. However, lesions that have received local treatment such as external-beam radiation therapy (EBRT) or radiofrequency ablation (RFA) must have progressed after these local treatment to count as measurable lesion
7. Participants with primary CNS tumors must meet all of the following criteria:

   1. Have received prior treatment including radiation and/or chemotherapy, as recommended or appropriate for the CNS tumor type
   2. Have >= 1 site of bi-dimensionally measurable disease (confirmed by magnetic resonance imaging (MRI) and evaluable by RANO criteria), with the size of at least one of the measurable lesions >= 1 cm in each dimension and noted on more than one imaging slice. Imaging study performed within 28 days before enrollment
   3. Must be neurologically stable based on neurologic exam at least for the last 7 days prior to enrollment. (based on medical examination/interview)
8. Corrected calcium <= 10.1 mg/dL
9. Phosphate <= 4.6 mg/dL
10. Required treatment washout period, from the last day of prior treatment until enrollment of this trial, is as follows:

    1. Antibody and other investigational drugs: >= 28 days
    2. Prior chemotherapy (excluding small-molecule targeted therapy), surgical therapy, radiation therapy: >= 21 days (>= 90 days from the date of the last radiation therapy for primary CNS tumors)
    3. Endocrine therapy, immunotherapy, small-molecule targeted therapy: >=14 days

Exclusion Criteria:

1. Participants with brain, subdural or leptomeningeal metastases
2. Participants with primary CNS tumor located in either cerebellum, brainstem, spinal cord, pituitary gland, optic nerve or olfactory nerve
3. Positive for either human immunodeficiency virus (HIV) antibody, HBs antigen, or HCV antibody (patients with positive HCV antibody but no detectable HCV-RNA are not excluded)
4. Negative for HBs antigen, but positive for HBs antibody or HBc antibody, and also positive for HBV-DNA quantification (not excluded if HBV-DNA is below detection sensitivity)
5. Child-Pugh score B or C
6. Participants with pericardial effusion, pleural effusion, or ascites requiring treatment
7. Have any of the following ocular diseases

   1. Grade 2 or higher corneal disorders
   2. Active retinopathy (e.g., age-related macular degeneration, central serous chorioretinal disease, retinal tear)
8. Participants whose toxicity of previous treatment has not recovered to Grade 1 or lower per Common Terminology Criteria for Adverse Events (CTCAE v5.0), except for alopecia, infertility, and the laboratory test results listed in the inclusion criteria
9. Participants who received a prior selective FGFR inhibitor in the recurrent/metastatic disease setting; except for patients with cholangiocarcinoma harboring FGFR2 fusion (Group D). Note that prior use of a multi-kinase inhibitor which includes anti-FGFR activity is acceptable after review by the lead investigator
10. Participants who need the use of drugs that strongly inhibits or induces the metabolizing enzyme cytochrome P450 (CYP) 3A
11. The presence of FGFR gatekeeper mutations as follows: FGFR1 V561, FGFR2 V564/565, FGFR3 V555/557, FGFR4 V550
12. The presence of any of the following coexisting driver gene abnormalities:

    1. Genetic mutations (excluding VUS): KRAS, NRAS, EGFR, or BRAF V600
    2. Gene translocations: ALK, ROS1, or NTRK

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Baseline up to 3.5 years
  Overall response rate (ORR) defined as the combined incidence of complete response (CR) and PR, confirmed no less than 4 weeks after the criteria for response are first met, based on RECIST v1.1. ORR will be confirmed by independent blinded central review assessment.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Baseline up to 3.5 years
  Overall response rate (ORR) defined as the combined incidence of complete response (CR) and PR, confirmed no less than 4 weeks after the criteria for response are first met, based on Response Assessment in Neuro-Oncology (RANO) criteria for primary Central Nervous System (CNS) tumor or RECIST v1.1 for other tumor type. ORR will be confirmed by local site investigator and/or independent blinded central review assessment.
Progression-free survival (PFS) | Baseline up to 3.5 years
  Progression-free survival (PFS) defined as the time from the date of enrollment to the date of the first documentation of objective progression of disease (PD), clinically diagnosed symptomatic deterioration, or death due to any cause in the absence of documented PD, whichever occurs first.
Overall Survival (OS) | Baseline up to 3.5 years
  Overall survival (OS) defined as the time from date of enrollment to date of death due to any cause.
Disease control rate (DCR) | Baseline up to 3.5 years
  Disease control rate (DCR) defined as the percentage of patients with a confirmed complete response (CR), partial response (PR) or stable disease (SD) as the best overall according to RECIST version 1.1.
Adverse event (AE) rate | From the first dose of the investigational product until 30 days after the last dose of study drugs
  Defined as the percentage of patients who experienced each adverse event. The severity of AEs were evaluated by the investigator according to Japan Clinical Oncology Group (JCOG) Japanese translation of the Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0-JCOG).
Adverse reaction (adverse drug reaction) rate | From the first dose of the investigational product until 30 days after the last dose of study drugs
  Defined as the percentage of patients who experienced each adverse reaction (causally related to the protocol treatment). The severity of AEs were evaluated by the investigator according to Japan Clinical Oncology Group (JCOG) Japanese translation of the Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0-JCOG).
Duration of response (DOR) | Baseline up to 3.5 years
  Duration of Response (DOR) defined as the time from the date of first documentation of CR or PR to the date of first documentation of disease progression or date of death from any cause, whichever occurs first.
Time to response (TTR) | Baseline up to 3.5 years
  Time to response (TTR) defined as the time from the date of first study dose to the date of first documentation of CR or PR according to RECIST version 1.1.

CONTACTS AND LOCATIONS:
Locations (7):
- Japan (7):
  - National Cancer Center Hospital, Chuo-ku, Tokyo, Japan
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Tohoku University Hospital, Aoba-ku, Sendai, Miyagi
  - Kyushu University Hospital, Higashi-Ku, Fukuoka
  - Hokkaido University Hospital, Kita-Ku, Sapporo, Hokkaido
  - Okayama University Hospital, Okayama
  - Kyoto University Hospital, Sakyo-ku, Kyoto

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chiba Y, Sudo K, Kojima Y, Okuma H, Kohsaka S, Machida R, Ichimura M, Anjo K, Kurishita K, Okita N, Nakamura K, Kinoshita I, Takahashi M, Matsubara J, Kusaba H, Yonemori K, Takahashi M. A multicenter investigator-initiated Phase 2 trial of E7090 in patients with advanced or recurrent solid tumor with fibroblast growth factor receptor (FGFR) gene alteration: FORTUNE trial. BMC Cancer. 2022 Aug 9;22(1):869. doi: 10.1186/s12885-022-09949-8. PMID 35945547